CLINICAL TRIAL: NCT00234962
Title: Factors Associated With Adherence in a Cohort of HIV Positive Subjects on a First Time PI Containing HAART Regimen: Observational Study of the Impact of Adherence on Viral Load for a HAART Regimen Containing Kaletra vs Other Selected PI Containing HAART.
Brief Title: Study of Adherence Effects and Clinical Outcomes of Kaletra Based HIV Antiviral Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUER-01-001
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: HIV Infection
Keywords: HIV Infection; HAART; Lopinavir; Ritonavir; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir

INTERVENTIONS:
Drug: Lopinavir/Ritonavir

SUMMARY:
The purpose of this study is to evaluate the effects of adherence on HIV antiviral response to treatment regimens containing Kaletra or other HIV protease inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Subject is documented HIV positive
* Subject is greater than or equal to 18 years of age.
* Subject currently on a regimen of either NNRTI + 2 Nucleoside Reverse Transcriptase Inhibitors NRTIs), two or three NRTIs who have failed regimen as evidenced by two consecutive viral loads with values over 1,000 copies/mL, the last one within the last three months, or
* Naïve subjects to ARV regimen who are required to begin a PI containing HAART regimen, or
* Subjects who have become intolerant to their current antiretroviral regimen and are required to be changed to a first time PI containing HAART regimen.
* Subject had laboratory testing within the previous three months and the most recent testing demonstrates all of the following: Hemoglobin >8.0 g/dL; Absolute neutrophil count >750 cells/mL; Platelet count >20,000/mL; ALT or AST <3 x Upper Limit of Normal (ULN); Creatinine <1.5 x ULN; Triglycerides <750 mg/dL.
* Subjects have no have evidence of grade III or IV adverse event or laboratory abnormality.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-08; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Antiviral efficacy by HIV RNA

SECONDARY OUTCOMES:
Treatment related discontinuations, predictors of adherence

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States